CLINICAL TRIAL: NCT04569370
Title: A Scoring System for Laparoscopic Cholycystectomy to Pick up Difficult Cases
Brief Title: A Scoring System for Difficult Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abobakr Mahfouz Abobakr, Resident Doctor, Assiut University
Other Study IDs: Scoring system for lap Choly
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Cholecystitis, Chronic
MeSH Terms: conditions — Cholecystitis; Bronchiolitis Obliterans Syndrome | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scoring Factor: Intervention: Procedure: Laparoscopic cholecystectomy
  Interventions: Procedure: Laparoscopic Cholecystectomy
- Difficult criteria: Intervention: Procedure: Laparoscopic cholecystectomy
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Surgical removal of Gall bladder using laparoscopy

SUMMARY:
Laparoscopic cholecystectomy is the treatment of choice for gall bladder stone disease. Difficult laparoscopic cholecystectomy (LC) is the most common "difficult" surgical procedure performed today, which possesses the potential to place the patient at significant operative risk.The aim of this study was to put a scoring system to avoid difficult laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Patients with symptomatic chronic calculous cholecystitis based on clinical and radiological correlation undergoing elective laparoscopic cholecystectomy at Assiut University hospitals will be included for the study of 100 patients will operated by single experienced laparoscopic surgeon.The scores are given on history, clinical examination and radiological findings one day prior to surgery on admission.

ELIGIBILITY:
Inclusion Criteria:

* Adults male and female age of or above 18 years
* Symptomatic chronic calculous cholecystitis
* Ultrasound confirmed Gall bladder stones

Exclusion Criteria:

* Complicated chronic calculous cholecystitis
* Malignant Gall bladder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with symptomatic chronic calculous cholecystitis based on clinical and radiological correlation undergoing elective laparoscopic cholecystectomy at Assiut University hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of preoperative scoring method for prediction of difficult laparoscopic cholecystectomy | 1 year
  Validation of sensitivity and specificity of Scoring system to predict difficulty of laparoscopic cholecystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Salah Ibrahim, Prof, Study Director — Professor at faculty of medicine

REFERENCES:
- [Background] Veerank N, Togale MD. VALIDATION OF A SCORING SYSTEM TO PREDICT DIFFICULT LAPAROSCOPIC CHOLECYSTECTOMY: A ONE-YEAR CROSS-SECTIONAL STUDY. J West Afr Coll Surg. 2018 Jan-Mar;8(1):23-39. PMID 30899702